CLINICAL TRIAL: NCT03810521
Title: A Phase I Dose-escalation Trial to Assess Safety and Efficacy of Cellistem-OA in Patients With Knee Osteoarthritis (CLT-OA1)
Brief Title: Dose-escalation of Cellistem-OA in Patients With Knee Osteoarthritis
Acronym: CLT-OA1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Francisco Espinoza, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLT-OA1
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis, Knee
Keywords: mesenchymal stromal cells
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CLT low-dose (Experimental): Umbilical cord derived-mesenchymal stromal cells at a dose of 2x10e6 cells / 3mL injected by an intra-articular infiltration of affected knee
  Interventions: Biological: umbilical cord derived-mesenchymal stromal cells
- CLT medium-dose (Experimental): Umbilical cord derived-mesenchymal stromal cells at a dose of 20x10e6 cells / 3mL injected by an intra-articular infiltration of affected knee
  Interventions: Biological: umbilical cord derived-mesenchymal stromal cells
- CLT high-dose (Experimental): Umbilical cord derived-mesenchymal stromal cells at a dose of 80x10e6 cells / 3mL injected by an intra-articular infiltration of affected knee
  Interventions: Biological: umbilical cord derived-mesenchymal stromal cells

INTERVENTIONS:
Biological: umbilical cord derived-mesenchymal stromal cells — Intra-articular infiltration of umbilical cord derived-mesenchymal stromal cells

SUMMARY:
A phase I dose-escalation trial to assess safety and efficacy of allogeneic MSC based-treatment (cellistem-OA) in patients with symptomatic knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Patient between 30 and 75 years old
* Knee-OA Kellgren Lawrence grade I to III
* Pain density according to visual analogue scale superior or equal to 50 mm
* Patelar condromalacia grade I to III
* Stable joint with normal physical exploration

Exclusion Criteria:

* Bilateral symptomatic disease
* Local or systemic infection
* Neoplasia
* Immunosuppression state
* Pregnancy
* Anticoagulant therapy
* Other types of arthritis
* Symptomatic disease of hip and/or spine
* Intra-articular infiltration with steroids in the last 3 months
* Intra-articular infiltration with hyaluronic acid in the last 12 months

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 months

SECONDARY OUTCOMES:
Change in WOMAC score | 6 months
Change in VAS score | 6 months
Changes in structural joint assessment by MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Espinoza, MD, Principal Investigator — CMO
Locations (1):
- Clínica Universidad de los Andes, Santiago, XIII, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matas J, Garcia C, Poblete D, Vernal R, Ortloff A, Luque-Campos N, Hidalgo Y, Cuenca J, Infante C, Cadiz MI, Khoury M, Luz-Crawford P, Espinoza F. A Phase I Dose-Escalation Clinical Trial to Assess the Safety and Efficacy of Umbilical Cord-Derived Mesenchymal Stromal Cells in Knee Osteoarthritis. Stem Cells Transl Med. 2024 Mar 15;13(3):193-203. doi: 10.1093/stcltm/szad088. PMID 38366909